CLINICAL TRIAL: NCT06102135
Title: To Evaluate the Acceptability (including Gastrointestinal Tolerance and Compliance) of an Adult Peptide 1.3 Kcal/ml Tube-feed Formula Containing Partially Hydrolysed Guar Gum (PHGG) Fibre.
Brief Title: Acceptability and Tolerance Study of Peptide Feed with Fibre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Peptide 003
Record Dates: First submitted 2023-08-22; First posted 2023-10-26 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2023-10

CONDITIONS: Dietary Exposure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients well established on tube feeds will act as their own control (Other): Patients in the control group will switch from current feed to new tube feed to assess tolerance and acceptability.
  Interventions: Dietary Supplement: Peptamen 1.3 PHGG

INTERVENTIONS:
Dietary Supplement: Peptamen 1.3 PHGG — The amount of tube feed will be assess by the health Care Professional.

SUMMARY:
Enterally fed adults with documented evidence of gastrointestinal intolerance will be recruited. Participants will be deemed by the investigator as having a clinical indication for enteral feeding with a fibre containing peptide formula. Data from 15 participants are required in order to submit an application to the Advisory Committee on Borderline Substances (ACBS) for product registration.

DETAILED DESCRIPTION:
To evaluate the acceptability (including gastrointestinal tolerance and compliance) of an adult enteral peptide formula containing Partially Hydrolysed Guar Gum (PHGG) fibre in 15 patients. This is a single arm, prospective, multi-centre study to evaluate the gastrointestinal tolerance and compliance over a fourteen-day period. Data will be collected using patient diaries to asses changes in GI tolerance and tube feed intake.

ELIGIBILITY:
Inclusion Criteria:

* Enterally fed adults feeding taking ≥60% of nutritional requirements from enteral nutrition

  * Patients with documented evidence of feeding intolerance or GI symptoms during enteral feeding, and who in the clinical judgement of the supervising dietitian may benefit from a peptide formula with fibre.
  * Aged 18 years and above.
  * Willingly given, written, informed consent from patient

Exclusion Criteria:

* Inability to comply with the study protocol, in the opinion of the investigator

  * Patients receiving mechanical ventilation, sedation or inotropic support
  * Patients on total parenteral nutrition
  * Known food allergies to any ingredients (see ingredients list) or galactosaemia
  * Patients with significant renal or hepatic impairment
  * Patients with planned changes to medication or treatments during the study period which may alter gastrointestinal function (e.g. chemotherapy). Changes in medications or nutritional products during the study intervention must be documented.
  * Participation in another interventional study within 2 weeks of this study.
  * Patients with a clinical indication for a low fibre or fibre free diet as advised by the healthcare team.
  * Patients with known or suspected ileus or mechanical bowel obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-09-05 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Assess tolerance via patient diaries | 14 days
  Daily assessment of diarrhoea, constipation, reflux, vomiting, wind, bloating
Daily formula intake | 14 days
  mL

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Wakefield, Principal Investigator — Newcastle Upon Tyne Hospital Trust; Nirouz Zarroug, Principal Investigator — Liverpool university Hospital Trust
Locations (2):
- United Kingdom (2):
  - Nutrition and Dietetics, Liverpool
  - Nutrition and Dietetics, Newcastle

IPD SHARING:
Plan to Share IPD: No
Will upload the data as it becomes available